CLINICAL TRIAL: NCT03567785
Title: Supporting Adherence to Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis: the Key to Successful Treatment Outcomes: the SUPIRIO-study
Brief Title: Supporting Adherence to Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis
Acronym: SUPIRIO
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Professor Wim Wuyts, Professor, Principal investigator, KU Leuven
Other Study IDs: S61427
Record Dates: First submitted 2018-05-09; First posted 2018-06-26 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis
Keywords: Therapy adherence
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is an irreversible, chronic and relentless lung disorder of unknown aetiology leading ultimately to respiratory insufficiency and death within 2-5 years after diagnosis. Treatment with the anti-fibrotic drug Pirfenidone slows down the disease progression and reduces the risk of acute exacerbations. Unfortunately, Pirfenidone represents a complex pharmacological regimen, in which patients have to take 3 tablets 3 times a day at mealtime. As for all chronically ill patients, adherence to a complex regimen might be challenging and nonadherence might reduce the full potential of Pirfenidone in patients with IPF. Due to extremely sparse availability of evidence on treatment adherence in the IPF population, it needs to be fully ascertained if, why, when and how many patients discontinue treatment or struggle to correctly take Pirfenidone as prescribed.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is an irreversible, chronic and relentless lung disorder of unknown aetiology characterised by a progressive destruction of lung parenchyma leading ultimately to respiratory insufficiency and death within 2-5 years after diagnosis. Treatment with the anti-fibrotic drug Pirfenidone slows down the disease progression and reduces the risk of acute exacerbations. Evidence also showed that treatment with Pirfenidone should be continued lifelong to maximise outcomes even in patients who experience disease progression during therapy. Unfortunately, Pirfenidone represents a complex pharmacological regimen, in which patients have to take 3 tablets 3 times a day at mealtime with a titration period in the first 3 weeks (i.e. 3 times 1 tablet of 267 mg during the first week, 3 times 2 tablets during the second week, and 3 times 3 tablets a week from week 3 onwards). As for all chronically ill patients, adherence to a complex regimen might be challenging and nonadherence might reduce the full potential of Pirfenidone in patients with IPF. Adherence is defined as "the extent to which a person' s behaviour - taking medication, following a diet, and/or executing lifestyle changes, corresponds with agreed recommendations from a health care provider"(WHO, 2003) and encompasses three phases namely, initiation, implementation and persistence.

Due to extremely sparse availability of evidence on treatment adherence in the IPF population, it needs to be fully ascertained if, why, when and how many patients discontinue treatment or struggle to correctly take Pirfenidone as prescribed. Furthermore, the investigators also don't know what the impact is of non-adherence to Pirfenidone on clinical outcomes in patients with IPF and whether good adherence is associated with a better health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IPF based on the 2011 ATS/ERS/JRS/LATA diagnostic criteria
* Patients who will start treatment with pirfenidone
* Patients of 18 years or older
* Oral fluency in Dutch or French
* Being able to provide written informed consent

Exclusion Criteria:

* Patients not managing their medications independently (e.g. Institutionalized patients, patients living in a nursing home or patients receiving homecare from a nurse). However, patients receiving help to prepare their medication from informal caregivers (i.e. family) are allowed to participate in the study.
* Patients not having their follow-up consultations at the University hospitals of Leuven.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with a recent diagnosis of IPF and starting on Pirfenidone at the University hospitals of Leuven will be invited to participate in the SUPIRIO study.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
The prevalence of non-adherence to pirfenidone (=non-initiation, discontinuation and non-implementation). | 1 year
  All patients included in the study will be equipped with a Medication Event Monitoring System (MEMS) (Aardex, Ch) to monitor the medication adherence continuously and to characterise adherence patterns. The MEMS bottle contains a cap which holds a microchip and a pressure-release system that records and stores the exact time and date each time the patient opens the bottle.The monitoring device will be read by the investigator using the MedAmigoTM platform. Patterns of medication intake will be analysed by the investigator.

SECONDARY OUTCOMES:
Impact of medication non-adherence on the forced vital capacity (FVC). | 1 year
  FVC data will be retrieved from the medical file of the patient.
Impact of medication non-adherence on progression-free survival. | 1 year
  Clinical data will be retrieved from the medical file of the patient.
Impact of medication non-adherence on quality of life measured with the EQ-5D-5L questionnaire. | 1 year
  Patients will receive the EQ-5D-5L measuring their health-related quality of life. The EQ-5D-5L is a standardised self-report questionnaire developed by the EuroQol group measuring the perceived health status of patients. It consists of the EQ descriptive system comprising five dimensions and the EQ visual analogue scale (VAS).
  Each dimension of the EQ descriptive system (i.e. mobility, self-care, usual activities, pain/discomfort, anxiety/depression) has 5 levels of response options (i.e. 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems and 5= extreme problems) and the combined answers of the dimensions result in a five-digit number describing the patient's health.
  Patients are also asked to fill in the EQ VAS where they have to report their current perceived health status on a vertical analogue scale. This scale ranges from 'best imaginable health state, i.e. 100' to 'worst imaginable health state, i.e. 0'.
Impact of health literacy on therapy adherence. | Baseline
  Health literacy will be assessed in this study because poor health literacy might be an important risk factor for therapy non-adherence and it was shown to be associated with a poorer capacity to comprehend and to follow medical advice as well as having poorer health outcomes. The self-administered single-item variant of the subjective health literacy screener (SHLS) will be given to the patients at baseline. In a validation study, the question 'how confident are you in filling out medical files by yourself' scored significantly better than two other investigated questions to detect patients with inadequate health literacy. This question will be scored on a 5-point likert scale (i.e. none, a little, some, most, all of the time), where a score between 0 and 2 (i.e. none, a little or some of the time) will be seen as inadequate health literacy.
Impact of depression on therapy adherence | 1 year
  The patient health questionnaire (PHQ-9) will be used to assess symptoms of depression, as it is a reliable and validated self-administered nine-item questionnaire based on the nine diagnostic criteria for DSM-IV depressive disorders. The score ranges between 0 and 27, since each item can be scored from 0 (not at all) to 3 (nearly every day). Cut-off points of 5, 10, 15, and 20 represent the lower limits of mild, moderate, moderately severe and severe depression, respectively.
Impact of barriers on therapy adherence | 1 year
  Barriers will be assessed with the adapted version of the 'immunosuppressive medication adherence barrier scale' (IMAB) developed by the transplant360 Task force. The questionnaire consists of 27 items that are scored on a 5-point likert scale (i.e. never, rarely, sometimes, often, always) resulting in a median score for all patients. Several barriers will be explored such as health beliefs, forgetfulness, disruption of the routine and complexity of the regimen.
Impact of medication non-adherence on quality of life measured with the K-BILD questionnaire. | 1 year
  Patients will receive the K-BILD questionnaire measuring their health-related quality of life. The K-BILD is a 15-item self-completed questionnaire measuring the health-related quality of life (HRQL) of patients with interstitial lung disease. It consists of three domains: breathlessness and activities, psychological and chest symptoms. Each question has a seven-point response scale resulting in a total score ranging between 0 and 100 with a higher score reflecting a higher HRQL.
Impact of medication non-adherence on quality of life measured with the SGRQ. | 1 year
  The St- George's Respiratory questionnaire (SGRQ) is a 50-item questionnaire consisting of two parts. The first part evaluates the symptoms (i.e. cough, sputum production, wheezing and breathlessness) and the second part evaluates the activities (i.e. activities causing breathlessness or limited by breathlessness) and the impacts (e.g. on employment, daily life, etc.). Each question is scored as positive (i.e. =1) or negative (i.e. =0) and the total score is expressed as a percentage where 0% represents the best possible health status and 100% the worst possible health status. A total score can be obtained as well as a score for each of the three components.
Impact of non-adherence on the diffusing capacity for carbon monoxide (DLco). | 1 year
  DLco data will be retrieved from the medical file of the patient.
Adherence to Pirfenidone | 1 year
  Patients will report their medication adherence by means of the validated Basel Adherence Assessment Scale for Immunosuppressive Medications (BAASIS). The questionnaire includes five questions about taking, dosing and timing of medication intake, as well as drug holidays, and treatment discontinuation. All deviating answers (i.e. questions answered by 'yes') will be defined as non-adherence.
Knowledge that patients have on their disease and treatment | 1 year
  Patients need to have the psychological capacity to adhere to their treatment meaning that they need to have adequate knowledge about their disease (e.g. severity of the disease) and treatment (e.g. side effects, dosing regimen). A specific questionnaire developed for this study will be given to patients to measure their knowledge about IPF and Pirfenidone. It consists of 6 true/false/I don't know questions on the treatment of IPF. Correct answers will receive a point resulting in a score ranging between 0 and 6 with higher scores reflecting a better knowledge.

OTHER OUTCOMES:
Adherence to limited alcohol intake | 1 year
  Patients are advised by the healthcare provider to limit their alcohol intake. Alcohol intake will be assessed using the AUDIT-C questionnaire. It consists of three questions with each five possible answers (i.e. a= 0 points, b= 1 point, c= 2 points, d= 3points and e= 4 points). A score of 4 or more in men and 3 or more in women is considered positive for identifying at risk drinking, defined as drinking at a level that might contain health risks.
Physical activity of patients | 1 year
  To measure the physical activity in this study, the two-item Brief Physical Activity Assessment Tool based on the physical activity guidelines, will be used. The total score ranges between 0 and 8 with a score of 4 or more reflecting an adequate physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Wuyts, Principal Investigator — Catholic University Leuven
Locations (1):
- University Hospitals Leuven, Leuven, BE, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delameillieure A, Dobbels F, Fieuws S, Leceuvre K, Vanderauwera S, Wuyts WA. Behavioural and psychological patterns of patients with idiopathic pulmonary fibrosis: a prospective study. Respir Res. 2022 May 14;23(1):124. doi: 10.1186/s12931-022-02041-6. PMID 35568881